CLINICAL TRIAL: NCT06127537
Title: Study on the Efficacy of Health Education and Therapeutic Group Factors on Cardiac Rehabilitation and Quality of Life in Coronary Patients
Brief Title: Study on the Efficacy of HE and Therapeutic Group Factors on CR and QoL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad de Extremadura (Other)
Collaborators: European Regional Development Fund (Other)
Responsible Party: Principal Investigator, Francisco Jose Rodriguez Velasco, Professor PhD, University of Extremadura, Universidad de Extremadura
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 134/2020; IB20186 (Other Grant/Funding Number: European Regional Development Fund); 134/2020 (Other: University of Extremadura Bioethics and Biosafety Committee); 19/10/2020 (Other: Research Ethics Committee - Extremadura Health Service)
Record Dates: First submitted 2023-09-27; First posted 2023-11-13 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Cardiac Rehabilitation
Keywords: Quality of Life; Cardiovascular Disease; Health Education
MeSH Terms: conditions — Cardiovascular Diseases; Health Education

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Health Education Programme in cardiac rehabilitation without a Therapeutic Intervention Group
- Experimental Group (Experimental): Health Education Programme in cardiac rehabilitation with a Therapeutic Intervention Group
  Interventions: Behavioral: Therapeutic Intervention Group

INTERVENTIONS:
Behavioral: Therapeutic Intervention Group — The therapeutic group factors that are worked on in the group session with a psychologist are:
  * Altruism.
  * Cohesion: feeling of belonging and acceptance in a group.
  * Universality: identification with the feelings, ideas or problems of the other group members.
  * Interpersonal-internalisation learning: the patient understands himself/herself by sharing his/her experience with the group.
  * Interpersonal-externalisation learning: the group offers the patient the possibility to express his own experience and to change his attitudes towards others.
  * Counselling.
  * Identification: assumption of behavioural patterns of other members as one's own.
  * Reactualisation of the family experience.
  * Understanding of one's own internal motivations.
  * Reciprocal stimulation: the improvement of other members encourages them to solve or approach their problems in a more favourable way.
  * Existential factors: empowerment of the individual.
  Arms: Experimental Group

SUMMARY:
This randomised study evaluates the efficacy of health education and therapeutic group factors on cardiac rehabilitation and quality of life in coronary patients attending cardiac rehabilitation programmes in Extremadura.

DETAILED DESCRIPTION:
Cardiac rehabilitation has been shown to be effective in improving the quality of life of patients who have suffered a cardiovascular event, as well as in preventing future cardiovascular events, demonstrating an increase in survival of between 20% and 30%, with a Class IA recommendation. Due to the prevalence of cardiovascular disease, both nationally and globally, it is important to study the benefits of these cardiac rehabilitation programmes in order to encourage their use. However, several studies have shown that for the programme to be effective, 5% to 10% weight loss must be achieved in patients, adequate nutritional education must be implemented, and behavioural and psychological intervention programmes must be incorporated in order to have an impact on adherence, psychological well-being, and coping with exercise intolerance. This project aims to study the effectiveness of health education and therapeutic group factors in cardiac rehabilitation and on quality of life in coronary patients in Cardiac Rehabilitation Units in Extremadura, including in the analysis anthropometric and body composition, nutritional, cognitive, emotional and lifestyle factors, which could act as mediators of cardiac function, reactivity to neuro-cardiovascular stress, anxiety, depression, anger-hostility, rehospitalisation, adherence, and adherence to treatment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of coronary heart disease, referred to the "Cardiac Prevention and Rehabilitation Unit".

Exclusion Criteria:

* Patients with disabling psychiatric disorders.
* Existence of pacemaker or automatic defibrillator.
* Presence of pregnancy or breastfeeding.
* Presence of medical conditions related to oncological conditions requiring chronic treatment with drugs or other substances.
* Any condition that, in the opinion of the investigators, would disqualify the subject from participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2024-01-31 (Estimated); Study Completion 2024-06-16 (Estimated)

PRIMARY OUTCOMES:
Changes in basal cardiac function and stress reactivity at 8 weeks | 0 and 8 weeks
  Changes in heart rate (bpm) are monitored at rest, during treadmill or stationary bicycle exercise and in recovery (by ergometry - PEG).
Changes in blood pressure over 8 weeks | 0 and 8 weeks
  Changes in blood pressure (mmHg) are monitored at rest, during exercise on a treadmill or stationary bike and in recovery. (by ergometry - PEG).
Change in cardiovascular health indicators over 8 weeks | 0 and 8 weeks
  Change in the Fuster-BEWAT score (FBS): this index is derived from cardiovascular health indicators blood pressure (mmHg), physical activity (METs), body mass index (kg/m2), fruit and vegetable consumption, and smoking status; 0-1 indicates poor cardiovascular health; 2-3, intermediate; and 4-5, ideal.
Changes in physical activity at 8 weeks | 0 and 8 weeks
  Changes in physical activity using the International Physical Activity Questionnaire (IPAQ): Weekly activity is recorded in Mets (Metabolic Task Equivalent or Metabolic Rate Units) per minute per week (Cat 1 - Low: <25 Mets / Cat 2 - Moderate: 25-600 Mets / Cat 3 - High: >1500 Mets).
Changes in maximum prehensile strength over 8 weeks | 0 and 8 weeks
  Changes in maximal upper limb prehensile strength by dynamometry (kg).
Changes in quality of life indicators over 8 weeks | 0 and 8 weeks
  Changes in the Spanish Quality of Life Questionnaire scores in post-infarction patients will be studied. The score per item ranges from 1 (never) to 5 (always). The minimum score is 40 (best health status) and the maximum 200 points (worst health status).
Changes in Physical Function quality score over 8 weeks | 0 and 8 weeks
  Items from the SF36 (Short Form 36) survey. The analysis of the responses is based on the calculation for domain with a scale between 0 (worst health status) and 100 (best health status), after coding, aggregation and transformation of the items that make up each domain.
Changes in Physical Role quality score over 8 weeks | 0 and 8 weeks
  Items from the SF36 (Short Form 36) survey. The analysis of the responses is based on the calculation for domain with a scale between 0 (worst health status) and 100 (best health status), after coding, aggregation and transformation of the items that make up each domain.
Changes in Bodily Pain quality score over 8 weeks | 0 and 8 weeks
  Items from the SF36 (Short Form 36) survey. The analysis of the responses is based on the calculation for domain with a scale between 0 (worst health status) and 100 (best health status), after coding, aggregation and transformation of the items that make up each domain.
Changes in General Health quality score over 8 weeks | 0 and 8 weeks
  Items from the SF36 (Short Form 36) survey. The analysis of the responses is based on the calculation for domain with a scale between 0 (worst health status) and 100 (best health status), after coding, aggregation and transformation of the items that make up each domain.
Changes in Vitality quality score over 8 weeks | 0 and 8 weeks
  Items from the SF36 (Short Form 36) survey. The analysis of the responses is based on the calculation for domain with a scale between 0 (worst health status) and 100 (best health status), after coding, aggregation and transformation of the items that make up each domain.
Changes in Social Function quality score over 8 weeks | 0 and 8 weeks
  Items from the SF36 (Short Form 36) survey. The analysis of the responses is based on the calculation for domain with a scale between 0 (worst health status) and 100 (best health status), after coding, aggregation and transformation of the items that make up each domain.
Changes in Emotional Role and Mental Health quality score over 8 weeks | 0 and 8 weeks
  Items from the SF36 (Short Form 36) survey. The analysis of the responses is based on the calculation for domain with a scale between 0 (worst health status) and 100 (best health status), after coding, aggregation and transformation of the items that make up each domain.
Changes in Health perception over 8 weeks | 0 and 8 weeks
  Changes in health perception will be calculated from the score of the Spanish Quality of Life Questionnaire in post-infarction patients. The score per item ranges from 1 (never) to 5 (always). The minimum score is 40 (best health status) and the maximum 200 points (worst health status).

SECONDARY OUTCOMES:
Changes in body weight composition over 8 weeks | 0 and 8 weeks
  Total patient weight are measured as a kilogram (kg).
Changes in body fat mass composition over 8 weeks | 0 and 8 weeks
  Total patient body fat mass are measured as a kilogram (kg).
Changes in body fat-free mass composition over 8 weeks | 0 and 8 weeks
  Total patient body fat-free mass are measured as a kilogram (kg).
Changes in estimated total body water composition over 8 weeks | 0 and 8 weeks
  Total patient estimated total body water are measured as a kilogram (kg).
Changes in protein composition over 8 weeks | 0 and 8 weeks
  Total patient protein are measured as a kilogram (kg).
Changes in bone mineral composition over 8 weeks | 0 and 8 weeks
  Total patient bone mineral are measured as a kilogram (kg).
Changes in Body Mass Index over 8 weeks | 0 and 8 weeks
  Weight (kg) and Height (m) will be combined to report BMI in kg/m^2.
Changes in CUN-BAE index over 8 weeks | 0 and 8 weeks
  CUN-BAE are calculated as -44.988+(0.503×age) +(10.689 ×sex) +(3.172×BMI) -(0.026×BMI2) +(0.181×BMI×sex) -(0.02×BMI×age) -(0.005×BMI2 ×sex) +(0.00021×BMI2×age), where male=0 and female=1 for sex, measuring age in years.
Changes in phase angle bioimpedance over 8 weeks | 0 and 8 weeks
  Phase angle is measured in degrees (º).
Changes in the percentage of carbohydrates ingested over 8 weeks | 0 and 8 weeks
  A standardised food consumption questionnaire will be used to assess dietary habits, which collects food intake over 7 days. The weekly nutrient intake will be transformed into "Food Composition Tables". The value obtained will be the percentage of carbohydrates (%).
Changes in the percentage of fat ingested over 8 weeks | 0 and 8 weeks
  A standardised food consumption questionnaire will be used to assess dietary habits, which collects food intake over 7 days. The weekly nutrient intake will be transformed into "Food Composition Tables". The value obtained will be the percentage of fat ingested (%).
Changes in the percentage of protein ingested over 8 weeks | 0 and 8 weeks
  A standardised food consumption questionnaire will be used to assess dietary habits, which collects food intake over 7 days. The weekly nutrient intake will be transformed into "Food Composition Tables". The value obtained will be the percentage of protein ingested (%).
Changes in the percentage of vitamins ingested over 8 weeks | 0 and 8 weeks
  A standardised food consumption questionnaire will be used to assess dietary habits, which collects food intake over 7 days. The weekly nutrient intake will be transformed into "Food Composition Tables". The value obtained will be the percentage of vitamins ingested (%).
Changes in kilocalorie intake over 8 weeks | 0 and 8 weeks
  A standardised food consumption questionnaire will be used to assess dietary habits, which collects food intake over 7 days. The weekly nutrient intake shall be transformed into "Food composition tables". The value obtained will be the number of kilocalories ingested (kcal).
Changes in adherence to the Mediterranean diet over 8 weeks | 0 and 8 weeks
  Changes in adherence to the Mediterranean diet. This will be studied using the Mediterranean Diet Adherence Questionnaire, which consists of 15 items with values ranging from <9 (low adherence) to >=9 (good adherence).
Changes in erythrocyte parameters over 8 weeks | 0 and 8 weeks
  Erythrocyte parameters are measured as a percentage [%]
Changes in glucose level over 8 weeks | 0 and 8 weeks
  Glucose is measured as a milligrams per decilitre [mg/dl]
Changes in plasma albumin parameters over 8 weeks | 0 and 8 weeks
  Plasma albumin are measured as a [g/dl]
Changes in total lymphocyte over 8 weeks | 0 and 8 weeks
  Total lymphocyte count are measured as a percentage [%]
Changes in total triglycerides levels over 8 weeks | 0 and 8 weeks
  Total lymphocyte count are measured as a milligrams per decilitre [mg/dl]
Changes in total cholesterol level over 8 weeks | 0 and 8 weeks
  Total cholesterol are measured as a milligrams per decilitre [mg/dl]
Changes in high-density lipoproteins levels over 8 weeks | 0 and 8 weeks
  High-density lipoproteins are measured as a milligrams per decilitre [mg/dl]
Changes in low-density lipoproteins levels over 8 weeks | 0 and 8 weeks
  Low-density lipoproteins are measured as a milligrams per decilitre [mg/dl]
Changes in psychological parameters over 8 weeks | 0 and 8 weeks
  Changes in STATE-TRAIT ANXIETY scores measured by the State-Trait Anxiety Questionnaire (STAI). It consists of 40 items divided into 2 subscales: trait and state, with Likert-type responses from 0 to 3. The score can range from 0 to 60. There are no cut-off points, but the direct scores are transformed into centiles according to sex and age.
Changes in adherence over 8 weeks | 0 and 8 weeks
  Change in Morisky Green Test scores. It consists of 4 items. The patient is considered to be compliant if he/she answers correctly to all 4 items. Parameter will be measured as compliant / not compliant-

CONTACTS AND LOCATIONS:
Overall Officials: Francisco J Rodríguez Velasco, PhD, Principal Investigator — University of Extremadura
Locations (1):
- Servicio Extremeño de Salud, Badajoz, Spain

IPD SHARING:
Plan to Share IPD: No